CLINICAL TRIAL: NCT04454827
Title: Fear of Hypoglycemia in Children and Adolecents With Type 1 Diabetes and Their Parents
Brief Title: Fear of Hypoglycemia in Children and Adolecents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Hypo-Fear-T1D-SI
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Type 1 Diabetes Mellitus; Fear of Hypoglycemia
Keywords: Type 1 Diabetes Mellitus; Fear of Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute symptoms of hypoglycemia influence all aspects of every day life and reduce quality of life of children and adolescents with type 1 diabetes and their parents. Encountering with hypoglycemia can result in fobic fear of low blood glucose levels in patients with type 1 diabetes and their parents.

DETAILED DESCRIPTION:
Fear of hypoglycemia is the most commonly reported problem in type 1 diabetes. By definition, hypoglycemia is a state of low blood glucose that is lower than 3,6 mmol/L. It can lead to uncomfortable counter-regulatory symptoms such as headaches, nervousness, weakness sweating, confusion, irritability, sleepiness and dizziness. In worst cases hypoglycemia can lead to loss of consciousness, seizures and death.

Unpredictability of episodes of hypoglycemia causes patients with diabetes and their family members to develop symptoms of anxiety and concerns related to hypoglycemia. The acute symptoms affect all fields of every day life and decrease quality of life of children and adolescents with type 1 diabetes and their parents. In some individuals and their families fear of hypoglycemia can lead to maintaining higher levels of blood glucose, excessive glucose monitoring, sleep deprivation, stress, obsessivity in self control, dependency to others etc.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than 0.5 year
* Age ≥ 1 year up to 25 years (inclusive)
* The subject/carer is willing to follow study specific instructions

Exclusion Criteria:

* Youth with maturity-onset diabetes of the young, hybrid, other, or missing type
* Any significant diseases / conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study
* Current use of the following medications: medications that are used to lower blood glucose such as Pramlintide, Metformin and GLP-1 analogs. Beta blockers, glucocorticoids and other medications, which in the judgment of the investigator would be a contraindication to participation in the study (Anticoagulant therapy e.g. Plavix, LMW heparin, Coumadin, Immunosuppressant therapy)

Ages: 1 Year to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents with type 1 diabetes and their parents
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Fear of Hypoglycemia | 5 months
  Questionnaires

SECONDARY OUTCOMES:
Time in ranges (below 3.9, 3.9-10, above 10 mmol/l | 1 year
  If available
HbA1c | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital Ljubljana, Ljubljana, Slovenija/Osrednja Regija, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided